CLINICAL TRIAL: NCT00155688
Title: A Genetic Linkage Study of Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 53ml; MH 59624-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 1998-12

CONDITIONS: Schizophrenia Sib-Pairs
Keywords: Schizophrenia; linkage; Taiwan; Han Chinese population
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
We propose to study 900 sib-pairs with the disorder. Our Specific Aims are: 1) To clinical assess a pedigree sample having adequate power to detect genes for schizophrenia. 2) To conduct a genome scan to find such loci. 3) To transmit all data to the NIMH designated cell repository and data management centers. We will attain these goals by achieving the following: 1) From Taiwan and China, we will collect 900 Han Chinese sib-pairs having DSM-IV schizophrenia. 2) We will examine all family members using the Diagnostic Interview for Genetic Study and the Family Interviews for Genetic Study. The PI participated in the development and field testing of these interviews and has an already established training program for their use. They have been translated into Mandarin by the Taiwanese investigators, who have used them in prior studies. 3) Blood samples will be sent to the NIMH designated cell repository for creation of lymphoblastoid cell lines. 4) Clinical Data will be entered using the database software created for the NIMH Human Genetics Initiative. Data will be vetted and sent to the NIMH designated data management center. 5) We will complete a genome scan using 450 markers spaced at an average of 10 cM intervals using markers that have been optimized for use in the Han Chinese population. The scan will be completed with no cost to the NIMH through an agreement with Millennim Pharmaceuticals, a biotechnogy company in the the Boston area that the PI has worked with on a prior genetic linkage study of schizophrenia. All genetic analyses will be approved by our consultant, Eric Lander, PhD. 6) All clinical data will be made available to the scientific community by the end of the funding period. All genotypes wil be available one year after they are created but no later than a year after the funding period. This project as feasible because 1) The PI has already coordinated one multi-site genetic linkage study of schizophrenia and has participated in a second. 2) We have a long-standing relationship with our Taiwanese collaborators and an effective, albeit, more recent working relationship with our Chinese collaborators. 3) We have conservatively estimated that each site has access to more than enough available families having two schizophrenic siblings. 4) The PI's Harvard team has had prior experience collaborating on genotyping and linkage analysis projects with Millennium Pharmaceuticals. This, and Millennium's prior genotyping experience shows that the genotyping phase of the work is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Han Chinese population
* Two Schizophrenia siblings, one normal parent and one normal sibling

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400
Dates: Start 1998-12; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University